CLINICAL TRIAL: NCT03767634
Title: Outcomes Following Early Parenteral Nutrition Use in Preterm Neonates
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4724
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-01

CONDITIONS: Neonatal Death; Prematurity
Keywords: Preterm neonate; Parenteral nutrition
MeSH Terms: conditions — Perinatal Death; Premature Birth; Hyperphagia | interventions — Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neonatal population (Project A): Neonates born between 1st January 2012 and 31st December 2017 and admitted to a neonatal unit in England, Scotland and Wales).
- No PN use (Project B): All neonates born between 30 and 33 weeks postmenstrual age in England, Wales and Scotland and admitted to a NHS neonatal unit between 1st January 2012 and 31st December 2017 who did not receive any parenteral nutrition (for any duration, by any intravenous route) in the first seven postnatal days.
- PN use (Project B): All neonates born between 30 and 33 weeks postmenstrual age in England, Wales and Scotland and admitted to a NHS neonatal unit between 1st January 2012 and 31st December 2017 who received any parenteral nutrition (for any duration, by any intravenous route) in the first seven postnatal days.
  Interventions: Other: Parenteral nutrition

INTERVENTIONS:
Other: Parenteral nutrition — Parenteral nutrition is the administration of an intravenous solution containing amino acids (with or without lipids) to provide nutritional support.
  Groups: PN use (Project B)

SUMMARY:
BACKGROUND

An essential part of neonatal care is providing nutrition to ensure that babies grow and develop. Providing this can be difficult in premature babies because their intestines are underdeveloped. They often have difficulty digesting milk so feeds are introduced gradually. To help babies grow and develop during this period, additional nutrition may be provided as a fluid into a vein; this is called "parenteral nutrition" (PN). Unfortunately, PN increases the risk of serious complications like bloodstream infection (also known as "sepsis"). For babies who are moderately premature there is little evidence to guide decision making about which babies will benefit from PN. This group of babies have more reserves of fat and are less dependent on PN, but are still at risk of sepsis. As a consequence, some doctors use PN and others do not.

AIMS

Firstly, to describe which babies are given PN during the first postnatal week in neonatal units in England, Scotland and Wales.

Secondly, to determine whether in babies born 7-10 weeks preterm (moderately premature), providing PN in the first week after birth, compared to not to providing PN, improves survival to discharge from the neonatal unit.

Finally, to evaluate if the early use of PN in moderately preterm babies affects other important outcomes in the neonatal core outcomes set.

IMPORTANCE

This work will describe the extent of PN use in England, Scotland and Wales. This is currently unknown. This project will improve understanding of the balance of benefits and harms of PN use in premature babies and will help doctors and parents make informed treatment choices.

METHODS

The investigators will use the National Neonatal Research Database (NNRD) to study all babies born in England, Scotland and Wales; they will identify which babies were given PN during the first week, and which were not. The investigators will use the NNRD to identify babies born 7-10 weeks prematurely and compare outcomes in babies that were given and not given PN in the first week after birth. The investigators will use statistical techniques to identify two sets of babies in the NNRD who are very similar (in terms of how prematurely they were born, their birth weight, and so on), the only difference being whether they were given PN or not. As the two groups will be similar any difference in their outcomes (such as survival) is likely to be due to whether or not they received PN.

DETAILED DESCRIPTION:
Premature birth abruptly ends the transplacental transmission of nutrients that allows normal foetal growth and development. Providing adequate nutrition is essential to allow premature babies to continue to grow and mature. Very preterm infants often have difficulty tolerating adequate volumes of milk feeds shortly after birth and so are given supplemental parenteral nutrition (PN). Preterm babies are among the highest PN users of all NHS patients. It has been estimated that PN is received by around 70% of neonatal unit admissions but it is not known exactly which babies receive PN. In addition, how PN affects outcomes has never been tested in a large scale, randomized, placebo controlled neonatal trial.

It is known that PN carries well established risks, of which the most serious and the most common is sepsis with estimates of risk ratios varying from 2.2 to 14.6. In addition there is a growing body of evidence that use of PN within the first seven days of admission to an intensive care unit is associated with worse outcomes in critically unwell adults and children. A subgroup analysis of the paediatric intensive care unit population focusing on neonates showed an increase in infections with early PN use. This suggests that uncertainty exists over the benefit of giving neonates PN in the early postnatal period. It is generally accepted that PN is beneficial to extremely preterm neonates, but in moderately preterm neonates the effect that PN use has on neonatal survival has never been conclusively demonstrated.

The uncertainty over how PN use affects neonatal outcomes is reflected by the wide variety in how PN is used in different units with large variation in use, timing and composition of PN. This is, in part, due to the lack of clear evidence of how PN affects neonatal outcomes like growth and survival. Neonates are also vulnerable to unanticipated treatment effects which can occur in different organ systems and so it is important to show that PN is not detrimental to important neonatal outcomes.

The postmenstrual age at which the nutritional benefits of PN outweigh the risks in moderately preterm babies (30-33 weeks postmenstrual age) is unknown. It is therefore unsurprising that their nutritional management is very variable. In moderately preterm neonates in 2012 and 2013 across England, Scotland and Wales PN was given to 45% of neonates, suggesting clinician equipoise around the balance of benefit to risk. Identifying whether moderately preterm neonates benefit from PN would have important implications for practice in the UK. This work will provide information to guide practice and inform future research.

In summary, PN is widely used in neonates but it is not known exactly how it is used in the UK. It is known to have risks and benefits but there is insufficient evidence to guide practice in moderately preterm neonates.

Study objectives:

* To describe the use of PN in neonatal units across England, Scotland and Wales.
* To identify if use of PN in the first seven postnatal days affects survival in neonates born between 30 and 33 weeks postmenstrual age.
* To explore how PN use in the first seven postnatal days affects other important neonatal outcomes in neonates born between 30 and 33 weeks postmenstrual age.

Study design:

Project A: an epidemiological survey of practice using the National Neonatal Research Database (NNRD).

Project B: a retrospective cohort study of matched groups of babies using data held in the NNRD.

ELIGIBILITY:
Inclusion Criteria:

Project A:

* Must be born between 1st January 2012 and 31st December 2017
* Must be admitted to a National Health Service (NHS) neonatal unit in England, Scotland or Wales

Project B:

* Must be born between 30 and 33 weeks postmenstrual age
* Must be born between 1st January 2012 and 31st December 2017
* Must be admitted to an NHS neonatal unit in England, Scotland or Wales

Exclusion Criteria:

Project A:

No exclusion criteria.

Project B:

* Major congenital gastrointestinal malformations
* Life limiting conditions
* Congenital conditions requiring surgery in the neonatal period
* Missing key background data (birthweight, sex or gestational age)
* Missing data for the primary outcome

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates born between 1st January 2012 and 31st December 2017 and admitted to a neonatal unit in England, Scotland and Wales).
Sampling Method: Probability Sample
Enrollment: 97507 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris RK Gale, PhD, Principal Investigator — Imperial College London
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Webbe J, Battersby C, Longford N, Oughham K, Uthaya S, Modi N, Gale C. Use of parenteral nutrition in the first postnatal week in England and Wales: an observational study using real-world data. BMJ Paediatr Open. 2022 Aug;6(1):e001543. doi: 10.1136/bmjpo-2022-001543. PMID 36053624
- [Derived] Webbe JWH, Longford N, Battersby C, Oughham K, Uthaya SN, Modi N, Gale C. Outcomes in relation to early parenteral nutrition use in preterm neonates born between 30 and 33 weeks' gestation: a propensity score matched observational study. Arch Dis Child Fetal Neonatal Ed. 2022 Mar;107(2):131-136. doi: 10.1136/archdischild-2021-321643. Epub 2021 Sep 21. PMID 34548324
- [Derived] Webbe J, Longford N, Uthaya S, Modi N, Gale C. Outcomes following early parenteral nutrition use in preterm neonates: protocol for an observational study. BMJ Open. 2019 Jul 9;9(7):e029065. doi: 10.1136/bmjopen-2019-029065. PMID 31289090

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Project A: 4,196,314 neonates were born in England and Wales. 347,959 neonates were admitted to NHS neonatal units . 62,147 neonates received PN during the first postnatal week.
  Project B: 37,302 neonates were born over the study period. 36,644 were admitted to an NHS neonatal unit.
  Prior to the propensity score analysis 843 neonates were excluded due to congenital conditions and 439 were excluded due to missing key data. This left 35,362 included in the propensity score analysis
Groups:
- Neonatal Population (Project A): Neonates born between 1st January 2012 and 31st December 2017 and admitted to a neonatal unit in England and Wales).
- No PN Use (Project B): All neonates born between 30 and 33 weeks postmenstrual age in England and Wales and admitted to a NHS neonatal unit between 1st January 2012 and 31st December 2017 who did not receive any parenteral nutrition (for any duration, by any intravenous route) in the first seven postnatal days.
- PN Use (Project B): All neonates born between 30 and 33 weeks postmenstrual age in England and Wales and admitted to a NHS neonatal unit between 1st January 2012 and 31st December 2017 who received any parenteral nutrition (for any duration, by any intravenous route) in the first seven postnatal days.
  Parenteral nutrition: Parenteral nutrition is the administration of an intravenous solution containing amino acids (with or without lipids) to provide nutritional support.
Period: Overall Study
Arm/Group | Neonatal Population (Project A) | No PN Use (Project B) | PN Use (Project B)
Started | 62145 | 19080 (8,146 neonates were included in the matched propensity score analysis) | 16282 (8,146 neonates were included in the matched propensity score analysis)
Completed | 62145 | 19080 (8,146 neonates were included in the matched propensity score analysis) | 16282 (8,146 neonates were included in the matched propensity score analysis)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neonatal Population (Project A) | No PN Use (Project B) | PN Use (Project B) | Total
Number analyzed (Participants) | 62145 | 8146 | 8146 | 78437
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62145 | 8146 | 8146 | 78437
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27965 | 3664 | 3733 | 35362
  Male | 34180 | 4482 | 4413 | 43075
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Use of Parenteral Nutrition (Project A)
Description: Any use of parenteral nutrition in the first seven days of postnatal life (assessed using daily data extracted from the National Neonatal Research Database as described in the project protocol)
  This outcome formed part of Project A ONLY, and in keeping with the research protocol is only analysed and reported for the babies in this research arm.
Time Frame: From birth until discharge home, assessed up to 1 year
Population: This outcome formed part of Project A ONLY, and in keeping with the research protocol has only been collected, analysed and reported for the neonates in this research arm. In Project B 'use of parenteral nutrition' formed a key background characteristic, and so this outcome is not reported for the two arms of Project B.
Measure: Count of Participants; unit: Participants
Arm/Group | Neonatal Population (Project A)
Number analyzed (Participants) | 347959
Participants | 62145

2. Primary Outcome: Survival to Discharge Home (Project B)
Description: Defined as recorded alive at final neonatal unit discharge
  This outcome formed part of Project B ONLY, and in keeping with the research protocol is only analysed and reported for the babies in this research arm.
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan This outcome formed part of Project B ONLY, and in keeping with the research protocol is only analysed and reported for the babies in this research arm.
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 7987 | 8057

3. Secondary Outcome: Late Onset Sepsis (Project B)
Description: Number of participants with diagnosed Later Onset Sepsis: defined in line with the Royal College of Paediatrics and Child Health National Neonatal Audit Programme (NNAP) definition "pure growth of a pathogen from blood" or "pure growth of a skin commensal" or a "mixed growth" after the first 72 hours of life
Time Frame: 72 hours of postnatal life to discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 59 | 179

4. Secondary Outcome: Necrotising Enterocolitis (Project B)
Description: Number of participants with diagnosed necrotising enterocolitis: defined using the NNAP definition: NEC may be diagnosed at surgery, post-mortem or on the basis of the following clinical and radiographic signs:
  At least one clinical feature from:
  (i) Bilious gastric aspirate or emesis (ii) Abdominal distension (iii) Occult or gross blood in stool (no fissure)
  And at least one radiographic feature from:
  (i) Pneumatosis (ii) Hepato-biliary gas (iii) Pneumoperitoneum
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Groups:
- PN Use (Project B): All neonates born between 30 and 33 weeks postmenstrual age in England and Wales admitted to a NHS neonatal unit between 1st January 2012 and 31st December 2017 who received any parenteral nutrition (for any duration, by any intravenous route) in the first seven postnatal days.
  Parenteral nutrition: Parenteral nutrition is the administration of an intravenous solution containing amino acids (with or without lipids) to provide nutritional support.
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 285 | 660

5. Secondary Outcome: Brain Injury on Imaging (Project B)
Description: Number of participants with diagnosed brain injury on imaging: defined as documented diagnosis of intraventricular haemorrhage (grade 3-4) or cystic periventricular leucomalacia
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 48 | 73

6. Secondary Outcome: Retinopathy of Prematurity (Project B)
Description: Number of participants with diagnosed retinopathy of prematurity: defined as a record of any retinopathy of prematurity on routine screening in the National Neonatal Dataset "retinopathy of prematurity ad-hoc form"
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 272 | 297

7. Secondary Outcome: Bronchopulmonary Dysplasia (Project B)
Description: Number of participants with diagnosed bronchopulmonary dysplasia: defined using the NNAP definition of significant bronchopulmonary dysplasia: Receiving respiratory support at 36 weeks corrected gestational age.
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 302 | 619

8. Secondary Outcome: Need for Surgical Procedures (Project B)
Description: Defined as any record of surgical procedure during the neonatal admission
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 69 | 147

9. Secondary Outcome: Seizures (Project B)
Description: Number of participants diagnosed as having a seizure: defined as any recorded diagnosis of seizures or seizure disorder
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Count of Participants; unit: Participants
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Participants | 81 | 114

10. Secondary Outcome: Weight (Project B)
Description: Weight z-score at discharge home. Weights at discharge home were converted to a z-score: a z-score of 0 represents the population mean, while score higher scores indicate a greater weight.
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Analysis of propensity score matched cohorts as per the pre-specified analysis plan
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 8146 | 8146
Z-score | 0.073 (0.98) | -0.024 (0.96)

11. Secondary Outcome: Head Circumference (Project B)
Description: Head circumference in centimetres at discharge; head circumference velocity (measured as increase in head circumference in centimetres/day) from birth until discharge
Time Frame: From birth until discharge home, assessed up to 1 year
Population: Initial analyses revealed considerable amounts of missing data (>90% missing): as the data represented under 10% of the true population it would not be possible to meaningfully summarise this data and it was highly unreliable (due to the high risk of systematic bias in this unrepresentative sample). For this reason full data relating to this outcome was not extracted from the National Neonatal Research Database as it was not in any way informative, and any further analysis was unjustified.
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Blindness (Project B)
Description: Defined as an answer of Yes to the question "Does this child have a visual impairment?" on the NNAP follow up form
Time Frame: From birth until two years of age
Population: as for outcome 11
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Deafness (Project B)
Description: Defined as an answer of Yes to the question "Does this child have a hearing impairment?" on the NNAP follow up form
Time Frame: From birth until two years of age
Population: as for outcome 11
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Ability to Walk (Project B)
Description: Defined as an answer of Yes to the question "Is this child unable to walk without assistance?" on the NNAP follow up form
Time Frame: From birth until two years of age
Population: as for outcome 11
Arm/Group | No PN Use (Project B) | PN Use (Project B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Project A: Adverse event data was not collected in this epidemiological study Project B: Adverse event data collected from birth until discharge home from hospital, assessed up to 1 year of age
Arm/Group | Neonatal Population (Project A) | No PN Use (Project B) | PN Use (Project B)
All-Cause Mortality (participants affected / at risk) | 5725/62145 | 163/8146 | 90/8146
Serious Adverse Events (participants affected / at risk) | 0/62145 | 0/8146 | 0/8146
Other Adverse Events (participants affected / at risk) | 0/62145 | 0/8146 | 0/8146

LIMITATIONS AND CAVEATS:
This study was a retrospective, observational study using data held within the National Neonatal Research Database.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03767634/Prot_SAP_000.pdf